CLINICAL TRIAL: NCT06932601
Title: The Validity of a Novel Diabetes Diagnostic Device and Its Feasibility as Metabolic Syndrome Diagnostic One. [TREARS STUDIES II]
Brief Title: Evaluation of a Novel Self-Sampling Earwax Tool for Chronic Disease Biomarkers [TREARS STUDIES II]
Acronym: Trears-II
Status: Not yet recruiting | Type: Observational
Sponsor: Trears (Industry)
Collaborators: Universidad del Desarrollo (Other); Hospital Padre Hurtado (Other)
Responsible Party: Sponsor
Other Study IDs: TREARS-II-2025-CL
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Syndrome; Diabetes; Hypertension; Obesity and Obesity-related Medical Conditions
Keywords: Trears; Earwax; Chronic Diseases; Long-Term & Continuous levels.; Self-Sampling Test
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Hypertension; Obesity; Chronic Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metabolic Syndrome Group: Participants with one or more diagnosed components of Metabolic Syndrome, such as hypertension, type 2 diabetes mellitus, dyslipidemia, or central obesity. No intervention is administered. Participants undergo non-invasive collection of earwax samples via a self-sampling device for sodium and other biomarker analysis. The aim is to assess the diagnostic value of earwax-based biomarkers compared with standard clinical reference measures.
- Healthy Control Group: Participants without any clinical diagnosis of metabolic syndrome or related chronic diseases. These individuals are used as baseline controls for comparison in the biomarker analysis. Earwax samples are collected using the same self-sampling method to evaluate sodium and other components. No treatment or intervention is provided.

SUMMARY:
Trears Biomarkers: A New Way to Manage Chronic Diseases

Trears Biomarkers are changing how we care for chronic diseases by focusing on patients' needs. People with chronic conditions often experience long-lasting changes in their bodies that typical tests do not accurately capture because they mostly measure short-term levels. These tests can be inconvenient, as patients frequently must travel to clinics, and some methods, like using needles, can be painful.

The Trears device, on the other hand, is easy and safe for people to use at home. It lets patients take their earwax samples, which they can send to the lab by regular mail, avoiding the hassle of mailing blood samples. This device could even make diagnosing diabetes more accurate.

Trears Biomarkers also investigates whether measuring sodium (salt) levels in earwax may be more reliable than a single blood pressure check and more straightforward than using a 24-hour blood pressure monitor. The aim is to enhance the diagnosis of all primary chronic conditions associated with Metabolic Syndrome (MetS), including diabetes, high cholesterol, obesity, and high blood pressure. These conditions are increasingly prevalent and already impact many people worldwide. With just one use, the Trears "multiplex" device could confirm a diagnosis typically requiring multiple tests.

Long-term lifestyle changes, like a healthy diet and regular exercise, work better than many drugs for treating MetS. Since the Trears device measures levels that change over time, it can give doctors a better picture of what's happening in a patient's body, allowing for more personalised recommendations. For instance, providing specific dietary advice could be more effective than simply prescribing medication, as it may lead to more lasting improvements in weight and blood pressure.

The device's design makes it accessible for home use, including by post, as earwax's natural bacteriostatic properties help preserve sample quality during mailing. In this study, we will test how effectively the Trears device works for diagnosing different types of diabetes and whether it can accurately track long-term levels of MetS markers. The device's new "multiplex" version might also support future point-of-care (POC) testing, allowing for the quick and convenient measurement of all MetS markers. We will consider how lifestyle factors - such as regular earplug use - might affect sample quality, ensuring the technology remains accurate and inclusive across diverse users. If necessary, we will introduce any potential changes in the Trears device design and/or marketing strategy after carefully considering feedback from our patients and their families, as outlined in Trears's mandate. Additionally, we will conduct an economic analysis to determine whether introducing the Trears device to a broader audience is financially sensible and essential. This will strengthen our position when launching our revolutionary technology in a conservative market.

DETAILED DESCRIPTION:
Title

The Validity of a Novel Diabetes Diagnostic Device and its Feasibility as Metabolic Syndrome Diagnostic One.

[TREARS STUDIES II] Herane-Vives, Andres1,2,3

1. Visiting Lecturer; Institute of Cognitive Neuroscience; Clinical, Educational & Health Psychology Department; Faculty of Brain Disease; University College London Alexandra House; 17-19 Queen Square; Bloomsbury; London; UK.
2. Visiting Lecturer; Affective Disorders Research Group, Centre for Affective Disorders, Department of Psychological Medicine, Institute of Psychiatry, Psychology & Neuroscience, King's College London, London, UK.
3. Trears Biomarkers Ltd, Founder & CEO, General Adult Psychiatrist Consultant, London, UK.

Abstract

Background: Long-term biomarker alterations feature chronic diseases. Metabolic Syndrome (MetS) is a cluster of them, i.e., diabetes, obesity, dyslipidaemia and high Blood Pressure (BP). Instead of genetic factors that could determine a categorical predisposition for this condition, MetS is primarily explained by the long-term effect of specific but dynamic lifestyles. Analysing MetS, as well as lifestyles, such as diet and physical activity, involves measuring long-term levels of many biomarkers. Because of their instant results, digital devices have been widely used for diagnosing MetS diseases, such as high BP, even though most can only record an "acute" level since, as with other chronic diseases, BP vary significantly over the short term. 24-hour sodium (Na+) could be used to reflect chronic blood pressure, considering its strong association with that variable at a population level. However, the "short-term" confounding effect of acute salt intake hinders its validity for reflecting chronic BP at the individual level. Otherwise, it would be more reliable than current devices, which are not only greatly affected by other "short-term" influences, such as acute stressors or "white coat" blood pressure but also time-consuming and impractical tests at a clinical level. Nonetheless, 24-h Na+ excretion showed that a more applied sample for accumulating Na+ should also be more effective at diagnosing this pandemic. A confounding role of "acute" salt intake over "chronic" Na+ levels could be avoided if the novel sample stored Na+ longer than urine. Trears Biomarkers' mission is to improve all chronic disease diagnoses. Trears device is the first self-sampling device for analysing earwax in the lab. It is an already patented medical device class I. Trears devices are as reliable as a popular clinical method (Reiner-Alexander syringe) for sampling earwax for analysis but more efficiently. Our previous Phase I study from TRL=6 to TRL=7/8 showed, when used, earwax was significantly better than gold-standard specimens, such as HbA1c from blood, for reflecting chronic levels of substances, which vary considerably over short-term, e.g., glucose. Trears devices can increase poor compliance among chronic patients, using annoying and time-consuming sampling methods, e.g. needles; reduce lab costs; and avoid stressful sampling methods that locally increase biomarkers' levels, which confuse their concentrations at a systemic level. Hypotheses: 1) It is expected that Trears device can improve glucose intolerance and diabetes diagnoses, and 2) it could also reflect other chronic disease biomarker concentrations, e.g. MetS ones, which are also variables over short-term, e.g., BP/Na+ and lipids such as cholesterol [HDL-C/LDL-C] and triglycerides [TD]. Objectives: This research will assess the sensibility and specificity of our device for diagnosing diabetes and glucose intolerance [Phase II study from TRL=7/8 to TRL=9], and 2] and its validity [new Phase I study from TRL=6 to TRL=7/8] for reflecting the average concentration of other chronic diseases biomarkers, such as MetS ones over 1- and 3 months. Methods: As earwax concentration does not differ between ear sides, the Trears Studies will be a longitudinal case [258]-control [258] study of four visits-screening and baseline visits and two follow-ups, one and two months apart. Novelty: From patients' homes and with single use, the Trears device could become the gold-standard diagnostic tool for diabetes and many other chronic conditions through this new Trears "multiplex" device, which could support the future development of the Trears multiplex Point-Of-Care [POC] test. Trears multiplex devices might finally enable the implementation of proper, precise measures for chronic disease patients.

Word count Abstract: 546 Main body: 11600

Keywords: Trears; Earwax; Self-Sampling Test; Chronic Diseases; POC; Long-Term & Continuous levels.

Background and Scientific and Technological Content

Trears Biomarkers aims to improve chronic disease diagnoses by measuring the long-term level of their diagnostic biomarkers using earwax samples, which patients themselves will take. This project covers two main areas:

Diagnostic, medical technology, and devices. Trears Biomarkers aims to continue validating its self-sampling device through its phase II study from TRL=7/8 to TRL=9, deep interviews, and health economic studies to confirm that the Trears device is the most reliable, affordable, and comfortable tool for screening, diagnosing, and following up different types of diabetes and glucose intolerance. The project will also test the device's stability under realistic mailing conditions, capitalising on earwax's bacteriostatic properties to support remote diagnostics.

Another focus of this project is developing another earwax self-sampling device, which can analyse many or "multiplex" chronic disease biomarkers. Trears Biomarkers market will move from the enormous but restricted diabetes testing market of 8.5 billion US dollars to enter the preventative health market constituted by healthy people, meaning soaring our original market size. That is why this project also aims to develop a single device (Trears Multiplex) which will accurately measure in the lab all biomarkers involved in a condition [MetS] featured by several comorbid chronic diseases, currently affecting between 20% and 30% of the US adult population [Phase 1 study from TRL=6 to TRL=7/8].

More than five years of work and solid scientific evidence support this revolutionary project, which ground-breaking aims to measure blood pressure using a single earwax sodium sample rather than a series of measurements done by unreliable sphygmomanometers or costly digital devices, e.g. Holter of BP.

To achieve these goals, this project includes:

A phase I & II prospective case-control study: 90 = +/- 7 days and will have four visits:

Screening (Day=-/+ 7),

Baseline (Day= 0), and two

Follow-ups 1 and

2, separated from the baseline by one (Day= 30) and two months (Day= 90), respectively.

Health economic analyses of different glucose and BP measurement methods for the diagnosis of diabetes/glucose intolerance and high BP, such as those taken by

Clinicians: plasma/serum from venous blood using syringes [Reference Test=4] and BP using sphygmomanometers [Reference Test=5].

Self-sampling methods, such as

i.- POCs use finger pricks (lancets) to measure biomarkers in situ from capillary blood [Reference Test=2], ii.- Continuous Glucose Monitoring [CGM] also in-situ but from the interstitial tissue, [Reference Test=3], iii.- Holter of BP, as approached measure to Continuous BP Monitoring [CBPM] [Reference Test=6] iv.- Home BP Monitoring [HBPM], as a manner to avoid "white coat" BP [Reference Test=7] and, v.- The Trears device uses earwax samples. [Reference Test=1]

A qualitative analysis of those sampling methods through deep interviews among a group of family doctors [GPs] and patients with diabetes or glucose intolerance, including perceptions of self-sampling feasibility and preferences regarding home mailing of biological samples, and,

Assess the validity of the Trears device in measuring chronic levels of MetS biomarkers to see whether it is worth developing a future Trears Multiplex POC Test.

At screening, participants will complete a short questionnaire on regular earplug use to allow stratified analysis of earwax composition and biomarker retention.

At baseline, a sub-study will test sample stability for postal transport by comparing bilateral earwax samples: one processed on-site during the day and the other mailed by the participant for delayed analysis (1, 3, or 7 days).

Problem and Opportunity

Non-Communicable Diseases (NCD) or chronic diseases, such as diabetes mellitus and MetS, constitute real pandemics. According to the National Health Contest in Chile, 12.3% of people over 15 had diabetes in 2017 (MINSAL, 2017). These figures indicate that our country has the most considerable prevalence of diabetes in South America (IDF, 2014). More outrageous is the figure which shows that the prevalence of a milder grade of hyperglycaemia or glucose intolerance (individuals with Impaired Glucose Tolerance [IGT] and Impaired Fasting Glucose [IFG] or diabetes) among Chileans adults is 36.0% (Nieto-Martinez et al., 2023). Furthermore, most all NCDs are chronic diseases. This explains several of their characteristics, such as the fact that long-term systemic alterations in different substances feature them. Indeed, a sustained elevation in glucose levels is mandatory for having diabetes (American Diabetes Association [ADA], 2010). However, current measurements from "short-term" specimens, such as serum, have significant limitations in the assessment of the average concentration of glucose level. Glucose levels also vary significantly during the day. Day-to-day hassles during periods of stress (Dagogo-Jack, 2010), smoking (Frati et al., 1996), high BP (Modan et al., 1985), Body Mass Index (BMI) (Hiller et al., 1998) and physical activity (Allen et al., 2009) can affect glucose levels. Some glucose measurements, such as fasting and postprandial glucose levels, have been standardised to provide a predictable glucose concentration level.

A single glucose test still does not accurately reflect the average concentration of glucose, which is the required level to monitor the glycaemic profile in metabolic chronic disorders such as diabetes (Makris & Spanou, 2011). These levels are usually found either below the mean, such as those seen when the Fasting Serum Glucose (FSG) level is taken, or below the average when Postprandial Serum Glucose (PSG) one is used (Peter et al., 2006). These blood samples need to be taken by clinicians, which increases their costs, apart from the fact that they can be associated with some side effects, such as local pain. Their analysis cost is high since these samples require specific transporting and storing conditions. A similar situation also ensues in another chronic disease, such as high BP. The devices used for measuring that variable only take a cross-sectional picture of it, a result that does not necessarily correlate with its chronic level, which is the biomarker needed for diagnosing this long-lasting condition. Furthermore, short-term levels of cholesterol and triglycerides, the other MetS biomarkers, also vary depending on caloric intake.

According to the World Economic Forum, treating chronic conditions such as diabetes and hypertension will cost 47 trillion dollars worldwide by 2030 (Gambert, 2024). In the U.S., 90% of health costs are associated with chronic conditions (CDC, 2024). Currently, the outcomes of these conditions could also be improved. Rather than being curative, available drugs are primarily symptomatic. Recent studies indicate that compared to those who engage in diet and physical activity, diabetic patients treated with hypoglycaemic drugs have poorer long-term outcomes, even though they may show lower Glycated Haemoglobin (HbA1c) levels (HC et al., 2008). This strongly suggests that medical interventions for chronic diseases need to have a sustained effect over time to be effective. Additionally, their impact should be monitored using a specimen (or device) capable of reflecting chronic glucose levels over the long term.

To complicate things more, chronic diseases are also comorbid conditions. Diseases such as diabetes, high BP, obesity, and dyslipidaemia are clustered in MetS. Then, medical interventions that use an integrative rather than a linear approach could be more effective for this group of conditions. They should also be tailored to each patient. A specific diet for someone who suffers from a MetS might be more effective at sustainably reducing weight and glucose levels over time than using two drugs, which can only impact those conditions acutely. Individual results, based on genotyping or gut microbiome tests, are currently compared with those obtained in the rest of the population, aiming to find inter-individual differences which support the design of standardised diets, such as energy-restricted with low salt or high sugar levels, among others. However, for most, their results have been poor, apart from those outlier cases of patients who suffer from a specific genetic alteration, e.g. congenital metabolic disorders, who benefit from a disease-orientated diet, which bans, for instance, a particular type of sugar. This approach for the design of different kinds of diets has been called personalised nutrition. Although highly effective in previous cases, the large variability seen in food responses, such as the postprandial plasma glucose responses -a common biomarker for chronic diseases- is primarily explained by intra- rather than inter-individual differences (Wolever, 2016). This reinforces the dynamic, rather than static, role of environmental factors (stressors) or lifestyles (physical activity levels) on food responses, as opposed to genetic factors.

Need or challenge

Chronic conditions mean chronic alterations, such as glycaemic and BP levels. Nonetheless, the samples or devices used for measuring their diagnostic biomarkers, such as blood or sphygmomanometers (or digital devices), are "short-term" ones, unable to average their levels over the long term and require clinicians or someone else to take the sample. Currently, HbA1c is the most used specimen to represent long-term glucose concentrations (Monnier et al., 2006; C. Rohlfing & Wiedmeyer, 2002). HbA1c is expensive to analyse and requires clinicians to take the sample. HbA1c is a form of haemoglobin showing a positive correlation with FSG and PSG. People without disease show weaker associations between HbA1c and fasting or postprandial glucose levels than diabetic patients (van 't Riet et al., 2010). This situation undermines the test's ability to screen a hyperglycaemic level amongst the general population (Dagogo-Jack, 2010).

Fasting glucose levels show stronger associations with HbA1c than postprandial glucose levels when measured in healthy people and diabetic patients with poor glycaemic control (Monnier et al., 2006); this means that HbA1c could be found within a healthy range in less severe diabetic patients who frequently have dietary transgressions. This limitation diminishes HbA1c's capacity to tightly monitor the mean glucose levels in glucose intolerance and mild diabetes. A more effective method for measuring the average concentration of glucose level should equally weigh its postprandial and fasting levels across the day. HbA1c measures the average plasma glucose concentration in the preceding three months. However, this glycated protein is more greatly weighted (75%) towards plasma glucose concentrations of the previous month (Leow, 2016). It is important to note that HbA1c does not provide predictable information about the glycaemic level over periods less than a month, such as those following changes (in weeks) after the prescription of hypoglycaemic drugs (Goldstein et al., 2004; K. J. Kim & Lee, 2012). It also has some additional limitations. HbA1c is not a precise method, as its levels can be affected by biological variables, such as age (Dagogo-Jack, 2010) or by common illnesses, such as anaemia (Sundaram et al., 2007) or several hemoglobinopathies (up to 7%) (Weatherall, 2011); even working long hours causes higher HbA1c levels (Azami et al., 2018).

HbA1c indirectly approximates the mean glucose level since it directly measures the protein rather than the sugar. Some authors even question the validity of HbA1c as a diagnostic test for diabetes mellitus and glucose intolerance due to the limitations above (Dagogo-Jack, 2010). Moreover, HbA1c can be an expensive and often inaccessible lab test in some developing countries (Sacks, 2011). This test requires a blood sample. Consequently, in contrast to self-sampling methods, the high cost of conventional sampling is tied to clinicians' work to collect the sample. Blood samples can have side effects, such as local infection and pain. Patients must travel to their healthcare providers to obtain venous blood, a procedure associated with local discomfort. This might explain why fewer than 40% of diabetic patients adhere to lab testing guidelines (Lian & Liang, 2014). Furthermore, current blood- or interstitial-based tests require strict cold-chain handling or in-person visits. Nonetheless, HbA1c remains one of the most requested lab tests yet is still underutilised (Salinas et al., 2012).

HbA1c, POC glucose, and HbA1c tests using capillary plasma have proven practical tools for self-monitoring these levels. As a CGM approach, a series of POC glucose tests has shown a strong association with HbA1c (C. L. Rohlfing et al., 2002a). However, POC glucose/HbA1c tests are not recommended for diagnosing diabetes due to significant variability among different brands and their lab-based results (A. I. Khan et al., 2006; Lenters-Westra & Slingerland, 2014). Indeed, the gold standard test for screening and diagnosing diabetes remains to measure glucose levels in the venous area rather than self-check tests or POC ones using capillary plasma. Furthermore, HbA1c lab-based results are not recommended as a screening test for milder hyperglycaemia or glucose intolerance. Therefore, diabetes and glucose intolerance diagnoses must still be confirmed using glucose testing, such as measuring glycemic levels two hours after the intake of a glucose load equivalent to 75 g of anhydrous glucose dissolved in water, also known as the Oral Glucose Tolerance Test (OGTT). The OGTT remains the gold-standard test for screening and diagnosing diabetes (WHO Press, 2006). However, the OGTT is a cumbersome, time-consuming, and expensive test. Olson et al. (2010) found that OGTTs revealed prediabetes in 35.8% and diabetes in 5.2%, whereas Hba1c provided Receiver Operating Characteristic (ROC) curve areas for diabetes of 0.79- 0.83, while ROC curve areas were ≤ 0.70 for dysglycemia or prediabetes. This discrepancy may be explained by milder degrees of hyperglycaemia that cannot oxidise HbA1c.

Later, CGM was developed to provide a method to track glucose levels throughout the day and night. CGM systems take glucose measurements at regular intervals, 24 hours a day, and translate the readings into dynamic data, generating glucose direction and rate of change (Mamkin et al., 2008). However, self-monitoring of blood glucose is still needed to inform treatment decisions in those using prandial insulin. There can be discrepancies between finger-stick blood glucose and sensor values. In addition to its increased cost, high and low glucose threshold alarms may be disruptive, and patients may develop 'alarm fatigue.' Information overload and the ability to make effective decisions about what to do with numbers and trends may be challenging for some patients (Klonoff et al., 2011; Walker et al., 2012). Overall, CGM may be a valuable educational and motivational tool for diabetes self-management, including using CGM. However, it also seems likely to be more time-consuming for patients and force them to focus on different aspects of diabetes, even though evidence suggests that they are reliable instruments for reflecting the average glycaemia in longer terms. Their most significant drawback is their delay in providing chronic glucose level results. Patients must wear CGM tests for the same length as the period prescribed to track, limiting their effectiveness. Still, wearing CGM devices, such as Free Style, for 14 days has been shown to provide a reasonable estimation of glucose metrics for three months as a measure of venous HbA1c in a large sample of type 1 diabetes patients with an R2 value of 0.84-0.86 for mean glucose, time at 70-180 mg/dL, and time>180 mg/dL, with lower values for time <70 mg/dL (0.76) and coefﬁcient of variation (0.70) (Riddlesworth et al., 2018). However, others found among children without diabetes that the same test, although correlated with post-OGTT glucose, had magnitude bias affecting fasting glucose and appeared to underestimate plasma glucose in those with overweight/obesity (Ghane et al., 2019), raising doubts about the validity of glucose measurements from interstitial tissue at reflecting the systemic glucose concentration. Regarding their correlation with HbA1c, previous studies have shown a discordance between the CGM and estimated average glucose derived by the conventional self-monitoring system with the standard laboratory HbA1c (M. L. Johnson et al., 2019). This is because OGTT and HbA1c differ intrinsically. HbA1c within an individual fluctuates a little daily, whereas an OGTT can reflect day-to-day differences in insulin secretion and action. As such, HbA1c reflects chronic glucose levels, whereas an OGTT reflects more acutely. Moreover, there is substantial interindividual variation in HbA1c at the same levels of glycemia (Nathan et al., 2008; C. L. Rohlfing et al., 2002b), so it is likely that short-term hyperglycaemic levels explained by OGTT have little impact on the level of HbA1c oxidation, which is what that lab test truly reflects. More recently, estimated HbA1c (eHbA1c) values have been calculated as HbA1c% = (mean glucose [MG] mmol/L + 2.59)/1.59 using CGM, e.g. Free Style for 14 days (Hill et al., 2011).

Poor compliance among high BP patients has been well-documented for decades, with fewer than 50% of these chronic patients returning for a medical checkup of that condition after a year (Engelland et al., 1979). Like CGM, a Holter is a non-invasive, ambulatory, continuous ECG monitoring device. The combined use of the Holter device alongside blood pressure (BP) monitoring has demonstrated advantages over traditional office BP measurements, particularly in providing numerous readings taken in the patient's daily environment (including during sleep). Additionally, it simultaneously and continuously records and stores ECG and blood pressure data for 24 hours, side by side, offering physicians more helpful information for evaluating the patient's cardiovascular status and detecting cardiac arrhythmias. This approach enhances the diagnostic value of the recorded data while increasing patient comfort and ease of use (Naser et al., 2022a). Kleinert et al. (1984) studied a sample of stable BP patients using a Holter device to measure BP continuously. It recorded their pressure with a cuff every 15 minutes while awake and every 30 minutes during sleep for 24 hours. They found a significant correlation between the mean BP readings taken by doctors and those recorded by patients themselves at home and in doctors' offices, using sphygmomanometers at regular intervals over the previous month.

Nevertheless, a single use of sphygmomanometers (Ali & Rouse, 2002) or digital tests (Nelson et al., 2008) are more practical (immediacy) for measuring BP, even though they are not very reliable since they can only measure "snapshots" of acute BP levels. Unlike self-sampling methods, which are immune to those confounders, their results are interrater, e.g., white coat hypertension, and interrater related when sphygmomanometers with different readers are used. Ultimately, nighttime BP and a non-dipper of nighttime BP are highly associated with mortality and cardiovascular events and provide better prognostic information than "office" BP (Kario & Williams, 2021), not reflected by most current devices requiring patients to be awake. Thus, a novel medical device for accurately measuring chronic BP should integrate the long-term impact of episodes of increased nocturnal BP while preventing the effect of short-term sodium covariates, such as salt intake transgressions. As expected, a similar situation also occurs with other MetS biomarkers. The postprandial peak of blood TG typically occurs 3-4 h after meal initiation (Lambert & Parks, 2012) or in the total, but not by subtype [HDL or LDL] cholesterol 2, as well 4 hours after having a meal (M. Kim et al., 2010).

Precision nutrition aims to develop tailored diets based on individual rather than genetic features, which can also vary depending on dynamic environmental rather than static genetic factors (Betts & Gonzalez, 2016). Most people would instead benefit from diverse diets, considering the dynamic impact of environmental factors on food responses. Betts and Gonzalez (2016) reinforced that point by saying that precise nutritional measures should be designed after considering the individual's baseline test results and then evaluating them using the individual's follow-up test results [test-retest]. Then, as opposed to personalised nutrition measures, precise ones can incorporate, at various points of the subject's lifespan, flexible amounts of that specific type of sugar that a personalised diet could only ban or allow since they are based on categorical genetic results. Thus, a future diagnostic and follow-up test for chronic diseases, such as the Mets, should be able to deliver chronic levels of all its biomarkers, such as cholesterol, High-Density Lipoprotein Cholesterol (HDL-C), Triglycerides [TG], glucose, and high BP in a single specimen to accurately track the impact of precise medical interventions for this condition over long-term. It should also be a safe and comfortable self-sampling test of low emission and production cost to avoid clinical work and polluting the environment. Trears Biomarker was born to improve the quality of life of chronic disease patients by making their conditions more likely to be monitored by our testing methods, whilst doctors can finally design more effective (precise) interventions at early stage (primary care) to avoid chronic disease progression.

State-of-the-Art Analysis

Background

Bees can accumulate substances through their honeycombs, and our wax can accumulate over the long term. Indeed, more than 60 years ago, Dr De Jorge became impressed with earwax's skills for accumulating substances, such as copper, despite their low systemic concentration (Jorge et al., 1964). Earwax's skills for reflecting chronic levels of different biomarkers were reinforced after observing that ceruminous (apocrine) glands, which produce this secretion, were not innervated (Bende, 1981). This means that they are immune to the effect of short-term variables, such as stress, food, and salt intake, among many other "acute" factors that hinder the use of "short-term" samples or devices for achieving the same goal. Earwax accumulates different biomarkers without being decomposed over time, allowing the posting of the sample without special shipping conditions, e.g., the cold chain needed, when "short-term" samples, such as blood, are used. As honeycombs, it possesses bacteriostatic properties, strengthening earwax's skills for accumulating different biomarkers. However, so far, no self-sampling device has shown to be as effective as the gold-standard clinical method, e.g., the Reiner-Alexander syringe for extracting impacted earwax, an external ear pathology. Indeed, cleaning earwax is not a medical indication. Despite that, cotton swabs are still the leading cause of eardrum perforation (Nussinovitch et al., 2004a). On the other hand, sampling earwax for analysis, if done by clinicians, would be an expensive procedure unlikely to become popular among the general population.

We have also included Na+ levels in earwax to be investigated in this study. Na+ and other elements have already been measured using earwax samples, finding, on average, 395.0 mEq/kg of Na+ in a sample of 22 participants, whereas, usually, the normal blood Na+ level fluctuates between 135 and 145 mEq/l. We are also interested in measuring earwax sodium because Na+ excretion over 24 hrs. is more reliable than a single BP measurement for determining chronic BP, although at the population level only, due to the confounding effect that acute salt intake plays in Na+ excretion over 24-hr. That lab test would still be unlikely

ELIGIBILITY:
Inclusion Criteria:

- i.People older than 35 years old ii.First-degree relative [parents or siblings] with diabetes. iii.Latin [Chilean] nationality iv.Women with a previous history of gestational diabetes or delivering a macrosomic (>9lb) baby v.Overweight or obese [BMI greater than or equal to 25 kg/m2] vi.Physical inactivity (no work-, transport-, or recreation-related physical activity in a typical week) vii.BP ≥130 and/or ≥80 mm Hg or use of antihypertensive medication viii.Self-reported diagnosis of prediabetes IFG, IGT or borderline diabetes. ix.Self-reported history of CVD: myocardial infarction, coronary heart disease, or stroke.

x.HDL-cholesterol < 35 mg/dL, triglycerides > 250 mg/dL, or lipid-lowering medication use xi.Women with polycystic ovarian syndrome xii.People with conditions associated with insulin resistance, such as acanthosis nigricansxiii.

Have non-alcoholic fatty liver disease.

Exclusion Criteria:

1. Participants with any ear disease, including external or internal otitis; Meniere syndrome or any form of dizziness; vertigo; malformation of the external ear; tinnitus; impacted earwax; current or previously perforated eardrums; individuals with tubes in their ears or who have had mastoid surgery; hearing loss or deafness, due to excess earwax production.
2. Asian ethnicity or intellectual disabilities due to their differences in the type and amount and type of earwax, respectively (Nussinovitch et al., 2004b; Pata et al., 2003).
3. This study will exclude people with very high blood glucose (blood sugar) levels [greater than or equal to 200 mg/dl] or with classic symptoms of high blood glucose.
4. Individuals with extreme ages under 18 years of age and over 75 years due to their different physiological responses and higher risk profiles.
5. Any conditions that might result in a significant change in glycemia, such as diseases requiring steroid therapy or pregnancy plans during the study period, will be exclusionary.
6. Any conditions that might result in a significant change in BP, such as diseases requiring steroid therapy or pregnancy plans during the study period, will be exclusionary.
7. Any conditions that might result in a significant change in BMI, such as plans for pregnancy during the study period, will be exclusionary.
8. Participants with hemoglobinopathies, anaemia, reticulocytosis, blood loss, transfusions, chronic renal or liver disease, high-dose vitamin C, or erythropoietin treatment (Nathan et al., 2007) will also be excluded (Nathan et al., 2007; Weatherall, 2011).
9. Individuals with a phobia of needles
10. Presence of infection or acute metabolic complications of diabetes, such as ketoacidosis or hyperosmolar state (coma).
11. Individuals with existing cardiovascular conditions (e.g., coronary artery disease, heart failure, arrhythmias) may be at increased risk of adverse events (e.g., arrhythmias, hypertensive crises) during salt and fat loading.
12. Individuals with morbid obesity (e.g., BMI > 40 kg/m²) if not safely manageable within the study protocols.
13. Current or heavy smokers, e.g. 20 or more cigarettes per day, due to the cardiovascular and metabolic impact of tobacco.
14. Individuals who abuse alcohol or any illicit substance due to their potential impact on liver and kidney function, electrolyte balance, and blood pressure regulation.
15. Participants adhering to strict dietary regimens (e.g., ketogenic diet, vegetarianism) may have atypical metabolic responses to high-fat and high-salt intake.
16. Individuals with existing renal diseases, e.g. Chronic Kidney Disease (CKD) stages 3-5 (eGFR <60 mL/min/1.73m²), history of acute kidney injury, nephrotic syndrome or significant proteinuria.
17. Individuals with recent illness or hospitalisation.
18. Current users of loop diuretics, thiazides, or potassium-sparing diuretics. insulin or oral hypoglycaemic agents, statins and other lipid-lowering drugs
19. Individuals with polypharmacy will also be excluded, including steroids or any medication that may affect sodium secretion and/or excretion in tablets, creams, or aerosols.
20. Allergy to medical grade adhesive or isopropyl alcohol used to prepare the skin.
21. Presence of skin lesions, scarring, redness, infection, or oedema at sensor application sites.
22. Individuals with Inflammatory Bowel Disease (Crohn's disease, ulcerative colitis), history of bariatric surgery within the past year, severe malabsorption syndromes, hepatitis, type 1 or Type 2 Diabetes Mellitus requiring insulin therapy, hyperaldosteronism or Addison's disease, thyroid disorders (e.g.,hyperthyroidism, hypothyroidism) not adequately controlled.
23. Use of non-steroidal anti-inflammatory drugs (NSAIDs) regularly.
24. The presence of any other condition is considered to warrant exclusion.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 to 75 years residing in Chile, recruited from Universidad del Desarrollo's primary care network, including Hospital Padre Hurtado and affiliated outpatient centers. The population includes individuals at risk for metabolic syndrome-defined by BMI ≥25 kg/m² and one or more ADA criteria risk factors-as well as healthy controls. Recruitment is stratified by earwax type and metabolic risk. No randomization will be applied
Sampling Method: Non-Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of self-sampled earwax glucose for diabetes and glucose intolerance detection | Baseline sampling with reference tests conducted within a ±5-day window
  This primary outcome assesses the sensitivity and specificity of self-sampled earwax glucose levels, measured in a central lab, in identifying individuals with diabetes and glucose intolerance. These will be compared against standard diagnostic methods including the Oral Glucose Tolerance Test (OGTT), HbA1c, capillary POC glucose, and Continuous Glucose Monitoring (CGM) across a 90-day period. Diagnostic performance metrics (sensitivity, specificity, PPV, NPV) will be calculated. The hypothesis is that earwax glucose will yield ≥85% sensitivity and ≥90% specificity compared to OGTT, with variability <5% and higher predictive accuracy than HbA1c.

SECONDARY OUTCOMES:
Correlation between earwax sodium concentration and chronic blood pressure | Single sampling at baseline; blood pressure history from past 3 months
  This outcome evaluates the relationship between self-collected earwax sodium concentrations and chronic blood pressure profiles. Earwax samples will be analyzed for sodium content and compared to standard ambulatory or home blood pressure monitoring values. The objective is to validate whether earwax sodium reflects long-term sodium intake and correlates with elevated or sustained blood pressure, distinguishing between normotensive, hypertensive, and salt-sensitive individuals. The hypothesis is that participants with hypertension will exhibit significantly higher sodium accumulation in earwax, with a correlation coefficient (r) ≥ 0.70.

OTHER OUTCOMES:
Correlation between earwax lipid concentrations (HDL, LDL, TG) and serum lipid profiles | Single sample collection with serum lipid panel obtained within ±5 days
  This outcome assesses whether lipids (HDL, LDL, triglycerides) measured in self-sampled earwax reflect standard serum lipid profiles in participants. Earwax samples will be analyzed in a central lab and compared with fasting lipid panels obtained within the same clinical visit. The hypothesis is that LDL and triglyceride concentrations in earwax will positively correlate with blood values (r ≥ 0.65), while HDL will show an inverse pattern. This will support the validity of earwax as a chronic lipid monitoring biospecimen, with relevance for Metabolic Syndrome diagnosis and monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Espinoza, B.Sc. M.D Msc. Ph.D., Study Chair — Pontificia Universidad Catolica de Chile

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) will not be shared publicly due to privacy concerns and regulatory restrictions under Chilean data protection laws. The data contains sensitive health and biometric information that could potentially identify participants, even in de-identified form. Additionally, the study is in an early exploratory phase and data will be used solely for internal analysis and validation purposes. Data sharing may be considered in future phases upon appropriate ethical and institutional review.

REFERENCES:
- [Background] Dedier J, Stampfer MJ, Hankinson SE, Willett WC, Speizer FE, Curhan GC. Nonnarcotic analgesic use and the risk of hypertension in US women. Hypertension. 2002 Nov;40(5):604-8; discussion 601-3. doi: 10.1161/01.hyp.0000035856.77718.da. PMID 12411450
- [Background] Gervitz LM, Nalbant D, Williams SC, Fowler JC. Adenosine-mediated activation of Akt/protein kinase B in the rat hippocampus in vitro and in vivo. Neurosci Lett. 2002 Aug 9;328(2):175-9. doi: 10.1016/s0304-3940(02)00495-0. PMID 12133582
- [Background] Halpern SD, Ubel PA, Caplan AL. Solid-organ transplantation in HIV-infected patients. N Engl J Med. 2002 Jul 25;347(4):284-7. doi: 10.1056/NEJMsb020632. No abstract available. PMID 12140307
- [Background] Lenters-Westra E, Slingerland RJ. Three of 7 hemoglobin A1c point-of-care instruments do not meet generally accepted analytical performance criteria. Clin Chem. 2014 Aug;60(8):1062-72. doi: 10.1373/clinchem.2014.224311. Epub 2014 May 27. PMID 24865164
- [Background] Khan NB, Thaver S, Govender SM. Self-ear cleaning practices and the associated risk of ear injuries and ear-related symptoms in a group of university students. J Public Health Afr. 2017 Dec 31;8(2):555. doi: 10.4081/jphia.2017.555. eCollection 2017 Dec 31. PMID 29456822
- [Background] Qiu Y, Yang J, Jiang W, Chen X, Bian C, Shi Q. A genomic survey on the immune differences among Sinocyclocheilus fishes. Commun Integr Biol. 2016 Nov 22;9(6):e1255833. doi: 10.1080/19420889.2016.1255833. eCollection 2016. PMID 28042381
- [Background] Nieto-Martinez R, Mechanick JI, Gonzalez-Rivas JP, Ugel E, Iglesias R, Clyne M, Grekin C. Revised Case Finding Protocol for Dysglycemia in Chile: A Call for Action in Other Populations. Endocr Pract. 2023 Aug;29(8):637-643. doi: 10.1016/j.eprac.2023.04.010. Epub 2023 Jun 1. PMID 37270107
- [Background] Chaliha C, Khullar V. Mixed incontinence. Urology. 2004 Mar;63(3 Suppl 1):51-7. doi: 10.1016/j.urology.2004.01.015. PMID 15013653
- [Background] Nathan DM, Kuenen J, Borg R, Zheng H, Schoenfeld D, Heine RJ; A1c-Derived Average Glucose Study Group. Translating the A1C assay into estimated average glucose values. Diabetes Care. 2008 Aug;31(8):1473-8. doi: 10.2337/dc08-0545. Epub 2008 Jun 7. PMID 18540046
- [Background] Zhang SW, Zhang YL, Pan Q, Cheng YM, Chou KC. Estimating residue evolutionary conservation by introducing von Neumann entropy and a novel gap-treating approach. Amino Acids. 2008 Aug;35(2):495-501. doi: 10.1007/s00726-007-0586-0. Epub 2007 Aug 21. PMID 17710364
- See also: Trears Studies II Project — https://youtu.be/Zf7T6szqAyw
- See also: Trears Device Instructions for Use — https://youtu.be/UfLzA80NwKQ